CLINICAL TRIAL: NCT00188669
Title: A Phase II Study of the Use of Pentoxifylline and a-Tocopherol in the Treatment of Chronic Breast Pain Associated With Breast Radiotherapy
Brief Title: The Use of Pentoxifylline and Vitamin E in the Treatment of Chronic Breast Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: date: August 2006. No annual renewal
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNH REB 02-0137-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Pentoxifylline; alpha-Tocopherol

INTERVENTIONS:
Drug: pentoxifylline
Drug: alpha-Tocopherol

SUMMARY:
An estimated 20 - 45 % of women treated with breast conserving treatment experience chronic pain in the treated breast. The aetiology of this is poorly understood. Some of these women have signs of chronic radiation mastitis. There is no accepted treatment for this condition. The combination of pentoxifylline and vitamin E has been shown to be effective in reversing radiation fibrosis in this region. Many of these patients have had a benefit in pain response in a time period of a few benefits. This study is a phase II study of these drugs for a 6 month trial period to assess the effect on chronic breast pain in breast cancer patients who are 3 months to 3 years post radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* UICC TNM stage 0 (i.e. in situ disease), 1 or 2 breast cancer patients treated with conservative surgery and adjuvant radiotherapy with chronic breast pain or tenderness, with or without fibrosis, within 3 months to 3 years following completion of radiotherapy
* Age 18 to 75 years of age
* Chronic symptoms localised to the breast treated with radiation, i.e. any one or more of the following- pain (not attributable to infection) or tenderness with or without associated oedema, fibrosis, necrosis or ulceration.
* Breast pain (maximum in the previous 24 hours) measurable on a Linear Analogue Scale with a length of 3cm or greater
* Prior treatment with radiation to the affected area i.e. in tangential breast fields or boost area
* Radiation completed at least 3 months and no longer than 3 years prior to study entry
* Informed consent

Exclusion Criteria:

* Active cellulitis in the breast
* Active malignant disease
* Any medical illness or condition judged likely by the local investigator to preclude safe administration of protocol treatment
* Contraindication to treatment with pentoxifylline (i.e. previously exhibited intolerance to pentoxifylline or other xanthines such as caffeine, theophylline or theobromine; recent cerebral and/or retinal haemorrhage; ischaemic heart disease; hypotension
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2002-07

PRIMARY OUTCOMES:
To assess improvement in breast pain with use of the interventional agents.
To assess improvement in patient function with the use of the interventional agents.

SECONDARY OUTCOMES:
To assess time to maximal improvement in pain, durability of response, quality of life changes during the study
To qualitatively characterise presenting pain syndromes
To examine techniques for objective assessment of breast edema and texture/fibrotic changes
To investigate the feasibility of the use of high resolution (40MHz) ultrasound and whether changes can be measured

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Levin, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada